CLINICAL TRIAL: NCT04133532
Title: Effect of Metoprolol in Post Alcohol Septal Ablation Patients With Hypertrophic Cardiomyopathy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Motol (Other)
Responsible Party: Principal Investigator, Hana Hnátová, medical doctor, resident in cardiology department, University Hospital, Motol
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HCMBB
Record Dates: First submitted 2019-10-16; First posted 2019-10-21 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Hypertrophic Cardiomyopathy
Keywords: Exercise tolerance; NTproBNP; Left ventricular outflow tract obstruction; Quality of life; Diastolic dysfunction
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic; Ventricular Outflow Obstruction, Left | interventions — Metoprolol

STUDY DESIGN:
Intervention Model Description: We will enroll 50 patients and divide them into two arms. Initially, arm A will be given metoprolol and arm B will not. We will evaluate the two groups after a sufficient time period (three months) and after that, patients will cross-over to the other treatment strategy for three months followed by a final evaluation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- metoprolol-no metoprolol (Experimental): After a washout period of one month following discontinuation of preceding beta-blocker medication patients will be given metoprolol 50 mg daily. The effect will be evaluated after three months of treatment. After that, another one-month washout period will commence followed by three months without metoprolol medication. Then, a final reevaluation will be performed.
  Interventions: Drug: Metoprolol
- no metoprolol-metoprol (Experimental): After a one-month washout period following discontinuation of preceding beta-blocker medication patients will continue another three months without a metoprolol medication. After that, an evaluation will be performed. Then they will be given metoprolol 50 mg daily for three months followed by a reevaluation.
  Interventions: Drug: Metoprolol

INTERVENTIONS:
Drug: Metoprolol — metoprolol 50 mg daily for three months

SUMMARY:
In this trial, the investigators will assess the effect of metoprolol in patients with hypertrophic cardiomyopathy who underwent alcohol septal ablation. The investigators will evaluate the quality of life, exercise tolerance, echocardiographic parameters and laboratory marker of heart failure and myocardial injury.

DETAILED DESCRIPTION:
In this trial, the investigators will assess the effect of metoprolol in patients with hypertrophic cardiomyopathy who underwent alcohol septal ablation.

The investigators will evaluate the quality of life, exercise tolerance, echocardiographic parameters and laboratory marker of heart failure and myocardial injury.

The investigators will enroll 50 patients that will meet all the inclusion criteria and will agree to participate in the trial. In patients with preceding beta-blocker medication, it will be discontinued and a washout period of one month will be provided. The investigators will assess baseline characteristics and then divide patients randomly into two arms based on their date of birth (even/odd days of the month).

Arm A will be given metoprolol 50 mg daily for three months, after this period the effect will be evaluated and metoprolol discontinued. A month-long washout period will follow and after an additional three months without metoprolol medication, patients will be reevaluated.

Arm B will be without metoprolol for three months and will be evaluated thereafter. Then the patients will be given metoprolol 50 mg daily for three months followed by a reevaluation.

The investigators will evaluate the effect of metoprolol by multiple methods at the end of the 5th and 9th months of the trial. Quality of life will be assessed by a questionnaire (The Kansas City Cardiomyopathy Questionnaire), exercise tolerance by a spiroergometry (VO2 max). A conventional echocardiographic examination and an examination focused on exercise-induced left ventricular outflow tract obstruction will be performed. The investigators will also measure NTproBNP from a blood sample as a laboratory marker of heart failure and high sensitive troponin as a marker of myocardial injury.

ELIGIBILITY:
Inclusion Criteria:

* Patients post alcohol septal ablation
* Pressure gradient in left ventricular outflow tract <30 mmHg
* Written consent to participate

Exclusion Criteria:

* History of atrial fibrillation
* Symptoms of Class III or IV of New York Heart Association functional classification
* Permanent pacemaker implant
* Age above 75

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2020-03-05 (Actual); Primary Completion 2023-02-23 (Actual); Study Completion 2023-02-23 (Actual)

PRIMARY OUTCOMES:
Change in exercise tolerance with and without metoprolol | At baseline, after three months of metoprolol medication, after three months without metoprolol medication
  VO2max during bicycle ergometer exercise test

SECONDARY OUTCOMES:
Change of quality of life with and without metoprolol: The Kansas City Cardiomyopathy Questionnaire | After three months of metoprolol medication, after three months without metoprolol medication
  The Kansas City Cardiomyopathy Questionnaire, score 0-100 (higher score means better outcome)
Change of concentration of biomarker of heart failure with and without metoprolol | After three months of metoprolol medication, after three months without metoprolol medication
  N-Terminal Pro-Brain Natriuretic Peptide concentration in blood sample
Change of concentration of a biomarker of myocardial injury with and without metoprolol | After three months of metoprolol medication, after three months without metoprolol medication
  High sensitivity troponin concentration in blood sample
Change in exercise induced pressure gradient in left ventricular outflow tract with and without metoprolol | After three months of metoprolol medication, after three months without metoprolol medication
  mmHg
Change in left ventricular diastolic function at rest with and without metoprolol | After three months of metoprolol medication, after three months without metoprolol medication
  Echocardiographic parameters of the transmitral flow and tissue Doppler

CONTACTS AND LOCATIONS:
Overall Officials: Josef Veselka, MD, PhD, Study Director — Motol University Hospital, Department of Cardiology
Locations (1):
- Motol University Hospital, Prague, Czech Republic, Czechia

REFERENCES:
- [Background] Gersh BJ, Maron BJ, Bonow RO, Dearani JA, Fifer MA, Link MS, Naidu SS, Nishimura RA, Ommen SR, Rakowski H, Seidman CE, Towbin JA, Udelson JE, Yancy CW; American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines; American Association for Thoracic Surgery; American Society of Echocardiography; American Society of Nuclear Cardiology; Heart Failure Society of America; Heart Rhythm Society; Society for Cardiovascular Angiography and Interventions; Society of Thoracic Surgeons. 2011 ACCF/AHA guideline for the diagnosis and treatment of hypertrophic cardiomyopathy: a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines. Circulation. 2011 Dec 13;124(24):e783-831. doi: 10.1161/CIR.0b013e318223e2bd. Epub 2011 Nov 8. No abstract available. PMID 22068434
- [Background] Maron BJ, McKenna WJ, Danielson GK, Kappenberger LJ, Kuhn HJ, Seidman CE, Shah PM, Spencer WH 3rd, Spirito P, Ten Cate FJ, Wigle ED; Task Force on Clinical Expert Consensus Documents. American College of Cardiology; Committee for Practice Guidelines. European Society of Cardiology. American College of Cardiology/European Society of Cardiology clinical expert consensus document on hypertrophic cardiomyopathy. A report of the American College of Cardiology Foundation Task Force on Clinical Expert Consensus Documents and the European Society of Cardiology Committee for Practice Guidelines. J Am Coll Cardiol. 2003 Nov 5;42(9):1687-713. doi: 10.1016/s0735-1097(03)00941-0. No abstract available. PMID 14607462
- [Background] HARRISON DC, BRAUNWALD E, GLICK G, MASON DT, CHIDSEY CA, ROSS J Jr. EFFECTS OF BETA ADRENERGIC BLOCKADE ON THE CIRCULATION WITH PARTICULAR REFERENCE TO OBSERVATIONS IN PATIENTS WITH HYPERTROPHIC SUBAORTIC STENOSIS. Circulation. 1964 Jan;29:84-98. doi: 10.1161/01.cir.29.1.84. No abstract available. PMID 14105035
- [Background] Cohen LS, Braunwald E. Amelioration of angina pectoris in idiopathic hypertrophic subaortic stenosis with beta-adrenergic blockade. Circulation. 1967 May;35(5):847-51. doi: 10.1161/01.cir.35.5.847. No abstract available. PMID 6067064
- [Background] Fananapazir L, Chang AC, Epstein SE, McAreavey D. Prognostic determinants in hypertrophic cardiomyopathy. Prospective evaluation of a therapeutic strategy based on clinical, Holter, hemodynamic, and electrophysiological findings. Circulation. 1992 Sep;86(3):730-40. doi: 10.1161/01.cir.86.3.730. PMID 1516184
- [Background] Gilligan DM, Chan WL, Joshi J, Clarke P, Fletcher A, Krikler S, Oakley CM. A double-blind, placebo-controlled crossover trial of nadolol and verapamil in mild and moderately symptomatic hypertrophic cardiomyopathy. J Am Coll Cardiol. 1993 Jun;21(7):1672-9. doi: 10.1016/0735-1097(93)90386-f. PMID 8496536
- [Background] Nistri S, Olivotto I, Maron MS, Ferrantini C, Coppini R, Grifoni C, Baldini K, Sgalambro A, Cecchi F, Maron BJ. beta Blockers for prevention of exercise-induced left ventricular outflow tract obstruction in patients with hypertrophic cardiomyopathy. Am J Cardiol. 2012 Sep 1;110(5):715-9. doi: 10.1016/j.amjcard.2012.04.051. Epub 2012 May 24. PMID 22633205
- [Background] Fifer MA, Vlahakes GJ. Management of symptoms in hypertrophic cardiomyopathy. Circulation. 2008 Jan 22;117(3):429-39. doi: 10.1161/CIRCULATIONAHA.107.694158. No abstract available. PMID 18212300
- [Background] Desai MY, Bhonsale A, Patel P, Naji P, Smedira NG, Thamilarasan M, Lytle BW, Lever HM. Exercise echocardiography in asymptomatic HCM: exercise capacity, and not LV outflow tract gradient predicts long-term outcomes. JACC Cardiovasc Imaging. 2014 Jan;7(1):26-36. doi: 10.1016/j.jcmg.2013.08.010. Epub 2013 Nov 27. PMID 24290569